CLINICAL TRIAL: NCT02428777
Title: Tramadol Versus Diclofenac for Prevention of Pain in Operative Outpatient Hysteroscopy: A Randomized Double Blind Placebo Controlled Trial
Brief Title: Tramadol Versus Diclofenac for Prevention of Pain in Operative Outpatient Hysteroscopy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdelGany Hassan, Lecturer of Gynecology and Obstetrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Hyst 5
Record Dates: First submitted 2015-04-24; First posted 2015-04-29 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Pain
Keywords: Hysteroscopy
MeSH Terms: conditions — Pain | interventions — Tramadol; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tramadol (Active Comparator): Women will receive oral tramadol 100 mg 1 hour before the procedure
  Interventions: Drug: Tramadol
- Diclofenac (Active Comparator): Women will receive oral diclofenac 100 mg 1 hour before the procedure
  Interventions: Drug: Diclofenac
- Placebo (Placebo Comparator): Women will receive an oral placebo 1 hour before the procedure
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tramadol — Women will receive oral tramadol 100 mg 1 hour before the procedure.
  Arms: Tramadol
Drug: Diclofenac — Women will receive oral diclofenac 100 mg 1 hour before the procedure
  Arms: Diclofenac
Drug: Placebo — Women will receive an oral placebo 1 hour before the procedure
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the effectiveness of Tramadol and diclofenac in reducing pain during operative outpatient hysteroscopy. Women undergoing operative hysteroscopy will be divided into 3 groups, the first group will receive Tramadol 100 mg 1 hour before the procedure, the second group will receive diclofenac 100mg 1 hour before the procedure and the third will receive a placebo. Pain will be assessed by a visual analogue scale

DETAILED DESCRIPTION:
Hysteroscopic examination is currently the most informative investigation for patients with abnormal uterine bleeding and infertility. Outpatient hysteroscopy involves the use of miniaturized endoscopic equipment to directly visualise the endometrial cavity, without the need of formal theatre facilities, general or regional anaesthesia.

Outpatient hysteroscopy is increasingly being used as a cost-effective alternative to in-patient hysteroscopy under general anaesthesia. Like other outpatient gynaecological procedures, however, it has the potential to cause pain severe enough for the procedure to be abandoned.

Opioid analgesics are widely used for the control of moderate to severe pain. Tramadol hydrochloride, a synthetic opioid is an orally active, clinically effective centrally acting analgesic having a lower incidence of respiratory depression, cardiac depression, side effects on smooth muscle and abuse potential as compared to typical opioid agents.

Diclofenac is a non steroidal anti inflammatory drug which inhibits the cyclooxygenase enzyme.

The study will be conducted in the outpatient hysteroscopy clinic in Cairo university hospitals. All patients attending the outpatient hysteroscopy clinic will be invited to participate in the study. The invitation will include a clear full explanation of the study and patients will provide oral consent. Written informed consent is not needed since the procedure and Patients will be included in the study if they give written consents.

Tramadol, diclofenac and placebo will be enclosed in sealed envelopes which will be numbered using computer generated random table. Neither the patient nor the physician will be aware of the drug used. 210 women will be categorized into 3 groups: Group I who will receive oral Tramadol 100mg (Trama®, Global Napi) orally 1 hour before the procedure, group II who will receive oral diclofenac 100mg (voltaren® 100, Novartis) 1 hour before the procedure, and group III who will receive an oral placebo.

Full history will be taken followed by general and local examination. The procedure will be done in the lithotomy position. Hysteroscopy will be done using a 5mm outer diameter continuous flow hysteroscope with a French working channel and a 30 degrees direction of view provided by Techno GmbH and CO. The hysteroscope will be introduced using the vaginoscopy technique, in which no speculum will be used. The cervix will be detected and the external os will be identified using the hysteroscope. The hysteroscope will be introduced in the uterine cavity. Saline will be used as the distension medium and the pressure will be set at 100mm Hg.

The anterior wall, posterior wall and tubal ostea will be visualised, any polyps, adhesions septa, congenital malformations or submucous fibroids will be noted. Endometrial biopsy will be taken using a semi-rigid, double action oval serrated biopsy forceps 40cm 5Charr provided by Tecchno medical GmbH. The used scissor will be a single action semi-rigid rounded tip scissors provided by Tecchno medical GmbH.

ELIGIBILITY:
Inclusion Criteria:

* Indication for operative outpatient hysteroscopy like endometrial biopsy, endometrial polyp, uterine septum, intrauterine adhesions, and loop retrieval.

Exclusion Criteria:

* Known allergy to tramadol or diclofenac.
* Diabetes, hypertension, gastritis, peptic ulcer, cardiac, renal or liver disease.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2015-04; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Pain during the procedure as measured by the visual analogue scale | 5 minutes after starting the procedure
  Women will be asked to score their pain using a visual analogue scale
Pain after the procedure as measured by the visual analogue scale | 30 minutes after completing the procedure
  Women will be asked to score their pain using a visual analogue scale

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - BeniSuef University hospitals, BeniSuef
  - Cairo university hospitals, Cairo

REFERENCES:
- [Background] Ahmad G, Attarbashi S, O'Flynn H, Watson AJ. Pain relief in office gynaecology: a systematic review and meta-analysis. Eur J Obstet Gynecol Reprod Biol. 2011 Mar;155(1):3-13. doi: 10.1016/j.ejogrb.2010.11.018. Epub 2011 Jan 20. PMID 21255900
- [Background] van Dongen H, de Kroon CD, Jacobi CE, Trimbos JB, Jansen FW. Diagnostic hysteroscopy in abnormal uterine bleeding: a systematic review and meta-analysis. BJOG. 2007 Jun;114(6):664-75. doi: 10.1111/j.1471-0528.2007.01326.x. PMID 17516956